CLINICAL TRIAL: NCT04778878
Title: Assessment of Chemotherapy-induced Peripheral Neurotoxicity Using a Point-of-care Nerve Conduction Study Device
Acronym: APPS
Status: Completed | Type: Observational
Sponsor: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Jussi Koivunen, Consultant, Oulu University Hospital
Other Study IDs: 48/2019
Record Dates: First submitted 2021-02-23; First posted 2021-03-03 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: CIPN, NCS
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mediracer® NCS — A point-of-care, hand-held nerve conduction device

SUMMARY:
The purpose of this study is to evaluate the feasibility of the Mediracer® NCS device in early detection of CIPN in patients receiving potentially neurotoxic substance (vincristine, oxaliplatin or docetaxel) as a part of their chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Planned initiation of oxaliplatin-, vincristine- or docetaxel-containing chemotherapy regimen [FOLFOX, XELOX, (R)-CHOP/CHOEP/CVOP, docetaxel, docetaxel-doxorubicin]
3. Age >18y
4. ECOG 0-2
5. Patient compliant with the study procedures

Exclusion Criteria:

1. Patient not fit/suitable for aforementioned chemotherapy regimen at baseline
2. Any prior postoperative or post-traumatic conditions affecting the sensory and/or motoric peripheral nerves
3. General vulnerability affecting the participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving neurotoxic chemotherapy (oxaliplatin, vincristine, or docetaxel) as cancer treatment.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Nerve conductivity | 6 weeks
  Nerve conductivity of n. medianus and ulnaris by Mediracer® NCS
Nerve conductivity | 12 weeks
  Nerve conductivity of n. medianus and ulnaris by Mediracer® NCS
Nerve conductivity | 18 weeks
  Nerve conductivity of n. medianus and ulnaris by Mediracer® NCS
Nerve conductivity | 24 weeks
  Nerve conductivity of n. medianus and ulnaris by Mediracer® NCS
Neuropathy related pain | 6 weeks
  Neuropathy related pain according to NPSI-assessment
Neuropathy related pain | 12 weeks
  Neuropathy related pain according to NPSI-assessment
Neuropathy related pain | 18 weeks
  Neuropathy related pain according to NPSI-assessment
Neuropathy related pain | 24 weeks
  Neuropathy related pain according to NPSI-assessment
Chemotherapy induced peripheral neuropathy (CIPN) | 6 weeks
  CIPN assessed by EORTC QLQ-CIPN20 questionnaire
Chemotherapy induced peripheral neuropathy (CIPN) | 12 weeks
  CIPN assessed by EORTC QLQ-CIPN20 questionnaire
Chemotherapy induced peripheral neuropathy (CIPN) | 18 weeks
  CIPN assessed by EORTC QLQ-CIPN20 questionnaire
Chemotherapy induced peripheral neuropathy (CIPN) | 24 weeks
  CIPN assessed by EORTC QLQ-CIPN20 questionnaire
Frequency of CIPN by CTCAE | 6 weeks
  Frequency of CIPN by CTCAE
Frequency of CIPN by CTCAE | 12 weeks
  Frequency of CIPN by CTCAE
Frequency of CIPN by CTCAE | 18 weeks
  Frequency of CIPN by CTCAE
Frequency of CIPN by CTCAE | 24 weeks
  Frequency of CIPN by CTCAE

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No